CLINICAL TRIAL: NCT05262088
Title: An Observational Cohort Study of Prognostic Value of Generalized Movements in the Diagnosis of Neurological Diseases in Children
Brief Title: Prognostic Value of Generalized Movements in the Diagnosis of Neurological Diseases in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West Kazakhstan Medical University (Other)
Responsible Party: Principal Investigator, Zhanna Zhussupova, PhD-doctoral, Department of Neurology, West Kazakhstan Medical University
Other Study IDs: 10.04.12.2020
Record Dates: First submitted 2022-02-16; First posted 2022-03-02 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy; Child Behavior Disorders; Neurologic Disorder; Pediatric Disorder
MeSH Terms: conditions — Cerebral Palsy; Child Behavior Disorders; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newborns: Assessment of the motor repertoire in children aged 0 to 5 months and its relationship with prenatal and perinatal factors and the results of neurological development in the second year of life.
  Interventions: Other: video recording of general movements

INTERVENTIONS:
Other: video recording of general movements — Video recording of general movements of children aged 3-5 days, then 4-5, 8-9, 12-13, 16-17, 20-22 weeks of life.
  At the age of 12 weeks of life, an assessment will be made on the Motor Optimality Scale (MOS).

SUMMARY:
To study of the evolution of general movements in children, to develop criteria for early diagnosis of neurological disorders to reduce early neurological disability.

It is observational longitudinal analytical cohort study.

DETAILED DESCRIPTION:
According to hypothesis, assessment of general movements is an early diagnostic tool for neurological disorders in children.

Combined estimates of epidemiological studies of neurological diseases in children under 3-5 years of age show that from 5.7% to 9.2% of children may have neurological disorders in different areas of development. According to the statistical report, the birth rate in the Aktobe region for 2019 and 2020 varies from 18.7 to 21.3 per 1000, that is, the expected birth rate in the Regional Perinatal Center of 7000-7500 newborns in 2021. The number of children in the region is 77360. Adjusted for an alpha error of 5% and a beta threshold of 20% (80% power), to achieve a predictive power of 0.95 and in accordance with selection criteria, expected 155 children with neurological disorders. Taking into account the cumulative frequency of disorders of neurological development of 9.2% in the study group, the sample should include 1800 children.

The present observational study is conducted in a population cohort of children of the Aktobe region. The motor repertoire of children aged 0 to 5 months will be evaluate and its relationship with demographic, prenatal, perinatal factors and the outcome of neurological development in the second year of life. The study (evaluation of general movements) is carried out by 3 specialists: the first specialist (the main researcher is a doctoral student) has access to all the survey materials, evaluates general movements from video materials, has an initial level of knowledge on the evaluation of general movements; 2 the specialist has a basic level (project manager) - has access to video recordings, has limited access to evaluate other variables; 3 the specialist has an expert level of knowledge (supervisor on a voluntary basis) on the evaluation of general movements, has access only to video recordings. As part of the pilot approach, all three specialists will evaluate the video recording of the movements of 50 infants, in the future it is planned to determine the reliability among evaluators using the Cohen's Kappa coefficient. Reliability will be considering high, when a coefficient of 0.61- 0.80 is reached.

The researcher on the 3rd-5th day of the child's life (home, hospital) explains in detail to parents the project being implemented. After receiving the informed consent of the parents, the researcher records the child's movements on video in accordance with the requirements, while simultaneously teaching the child's mother.

At the first stage, all full-term newborns will be examined. The examination is carried out no earlier than 3 days (adaptation period) after birth. At this stage, the child's general condition and neurological status will be assessed. Clinical data include the status of breastfeeding and the health status of the baby from the moment of birth. The Apgar scale will be used to assess the general condition of the newborn. In the presence of perinatal asphyxia, indicators on the Sarnat scale for neonatal encephalopathy will be used. Neonatal encephalopathy, acute encephalopathy and/or hypoxic-ischemic encephalopathy will be evaluated according to clinical and laboratory criteria. The following data will be evaluated: the sex of the baby, the age of the baby in days, a family member with a disability, the gestational age of the child at birth, birth weight, head circumference, the nutritional status of the baby (breast, artificial, mixed). These variables, except for the latter, are continuous (quantitative) indicators, all other data will be categorical. The weight and circumference of the child's head will be considered a pathology if the deviation is more than 2 standard deviations (SD) below the median (according to WHO). All data is entered into a specially designed individual registration card.

At the next stage, general movements are evaluated in the following age periods: 3-5 days, 4-5, 8-9, 12-13, 16-17, 20-22 weeks of life. The division into stages of assessment is fundamental, in the period from birth to 8-9 weeks, general movements are evaluated, which are classified as normal, abnormal or cramped synchronized. Normal general movements include an oscillating sequence of movements of the arms, neck, torso and legs. They increase and decrease with changes in intensity, speed and range of motion. Their beginning and end are usually gradual and smooth. The change of direction and rotation along the axes of the trunk and limbs is smooth and elegant. Abnormal movements will be the following movements: "poor repertoire" - the sequence of movements, their intensity, speed and range of movements are not changeable; "cramped synchronized" - the muscles of the trunk and limbs seem stiff and contract almost simultaneously, and then relax almost simultaneously.

The researcher on the 3rd-5th day of the child's life (home, hospital) explains in detail to parents the project being implemented. After receiving the informed consent of the parents, the researcher records the child's movements on video in accordance with the requirements, while simultaneously teaching the child's mother.

At the first stage, all full-term newborns will be examined. The examination is carried out no earlier than 3 days (adaptation period) after birth. At this stage, the child's general condition and neurological status will be assessed. Clinical data include the status of breastfeeding and the health status of the baby from the moment of birth. The Apgar scale will be used to assess the general condition of the newborn. In the presence of perinatal asphyxia, Sarnat scale for neonatal encephalopathy will be used. Neonatal encephalopathy, acute encephalopathy and/or hypoxic-ischemic encephalopathy will be evaluated according to clinical and laboratory criteria. The following data will be evaluated: the sex of the baby, the age of the baby in days, a family member with a disability, the gestational age of the child at birth, birth weight, head circumference, the nutritional status of the baby (breast, artificial, mixed). These variables, except for the latter, are continuous (quantitative) indicators, all other data will be categorical. The weight and circumference of the child's head will be considered a pathology if the deviation is more than 2 SD (standard deviations) below the median (according to WHO). All data is entered into a specially designed individual registration card.

At the next stage, general movements are evaluated in the following age periods: 3-5 days, 4-5, 8-9, 12-13, 16-17, 20-22 weeks of life. The division into stages of assessment is fundamental, in the period from birth to 8-9 weeks, general movements are evaluated, which are classified as normal, abnormal or cramped synchronized. Normal general movements include an oscillating sequence of movements of the arms, neck, torso and legs. They increase and decrease with changes in intensity, speed and range of motion. Their beginning and end are usually gradual and smooth. The change of direction and rotation along the axes of the trunk and limbs is smooth and elegant. Abnormal movements will be the following movements: "poor repertoire" - the sequence of movements, their intensity, speed and range of movements are not changeable; "cramped synchronized" - the muscles of the trunk and limbs seem stiff and contract almost simultaneously, and then relax almost simultaneously.

The obtained data will be entered into a special scheme with the subsequent construction of the trajectory of changes for the analysis of the evolution of general movements.

General movements will be recorded on a 5-minute video. The video is shot from above the baby (with the capture of the whole body of the child) lying on his back, in the conditions of the maximum absence of sensory and tactile stimulation. At the same time, the child should be awake, not hungry and lightly dressed. The videography technique is not complicated, does not have strict training criteria, can be carried out by parents, medical staff.

In the catamnestic observation of children, the neurological status at the age of 1, 2, 5, 12, 18 and 24 months of life will bee assess. Neurological status is assessed according to the Hammersmith Infant Neurological Examination (HINE) scale. This method is easy to use and was developed for the examination of children aged 2 to 24 months. It includes 26 items that evaluate the function of cranial nerves, posture, quality and quantity of movements, muscle tone, reflexes and reactions. Each item is rated from 0 (minimum) to 3 (maximum score), which gives a total score from 0 to 78. Sensitivity and specificity are about 0.90. According to this scale, the child's posture and posture are evaluated.

According to the results of the neurological examination, 2 groups will be identified: healthy and neurological disorders, which may include motor disorders associated with cerebral palsy, motor disorders not associated with cerebral palsy, epilepsy, orthopedic congenital malformations, muscular dystrophy, spinal muscular atrophy, developmental delay, genetic disorders, visual impairment, hearing impairment or a high risk of mental disorders.

Children with manifestations of abnormal movements, up to 5 months of age, all will undergo neurosonography (NSG - ultrasound of the brain).

Verification of the clinical diagnosis will be carry out according to the diagnostic criteria of the current clinical protocols of the Ministry of Health of the Republic of Kazakhstan and international classifications. In addition, all data will be entering into special designed individual registration card (IRC).

ELIGIBILITY:
Inclusion Criteria:

* all full-term newborn children born in the city of Aktobe in the period from
* both male and female children
* patients whose parents have signed an informed consent to data collection
* patients, as long as parents are able to comply with the requirements of the study protocol.

Exclusion Criteria:

* premature babies
* children with suspected chromosomal and metabolic diseases
* children of parents who have not signed the informed consent.
* children with fatal outcome are excluded in dynamics

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The present observational study is conducted in a population cohort of children aged 0 to 5 months of life. The motor repertoire of children aged 0 to 5 months will be evaluate, and its relationship with demographic, prenatal, perinatal factors and the results of neurological development in the second year of life. Newborn boys and girls are included in the study with the informed consent of their parents.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Changing the frequency of disability of children with neurological disorders | 2 years
  Early diagnosis of neurological disorders, and early rehabilitation interventions

CONTACTS AND LOCATIONS:
Overall Officials: Dinmuhammed Ayaganov, Principal Investigator — West Kazakhstan Medical University
Locations (1):
- Zhanna Zhussupova, Aktobe, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Einspieler C, Bos AF, Krieber-Tomantschger M, Alvarado E, Barbosa VM, Bertoncelli N, Burger M, Chorna O, Del Secco S, DeRegnier RA, Huning B, Ko J, Lucaccioni L, Maeda T, Marchi V, Martin E, Morgan C, Mutlu A, Nogolova A, Pansy J, Peyton C, Pokorny FB, Prinsloo LR, Ricci E, Saini L, Scheuchenegger A, Silva CRD, Soloveichick M, Spittle AJ, Toldo M, Utsch F, van Zyl J, Vinals C, Wang J, Yang H, Yardimci-Lokmanoglu BN, Cioni G, Ferrari F, Guzzetta A, Marschik PB. Cerebral Palsy: Early Markers of Clinical Phenotype and Functional Outcome. J Clin Med. 2019 Oct 4;8(10):1616. doi: 10.3390/jcm8101616. PMID 31590221
- [Result] Toldo M, Varishthananda S, Einspieler C, Tripathi N, Singh A, Verma SK, Vishwakarma K, Zhang D, Dwivedi A, Gupta R, Karn S, Kerketta N, Narayan R, Nikam Singh K, Rani S, Singh A, Singh D, Singh KP, Singh N, Singh N, Singh R, Singh SP, Srivastava R, Srivastava S, Srivastava S, Yadav G, Yadav P, Yadav S, Yadav S, Marschik PB. Enhancing early detection of neurological and developmental disorders and provision of intervention in low-resource settings in Uttar Pradesh, India: study protocol of the G.A.N.E.S.H. programme. BMJ Open. 2020 Nov 3;10(11):e037335. doi: 10.1136/bmjopen-2020-037335. PMID 33148727